CLINICAL TRIAL: NCT06355986
Title: Community-Based, Cluster-Randomized Trial of Electronic Alert-Based Computerized Decision Support to Prevent Stroke in High-Risk Ambulatory Patients With Atrial Fibrillation (AF-ALERT3)
Brief Title: Computerized Decision Support to Prevent Stroke in Atrial Fibrillation
Acronym: AF-ALERT3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Staff Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 39039039AFL4016
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; stroke; prevention; computerized decision support; anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Intervention Model Description: 2500-patient U.S. multicenter, community-based Quality Improvement Initiative in the form of a cluster-randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assignment to a particular cluster (ALERT or NO ALERT) will be masked to the patient participant, investigator, and outcomes assessor. Since the intervention is a computer alert to the provider of record, he/she will be aware of whether or not a notification is provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert (Experimental): For Alert cluster sites, an on-screen electronic alert will be issued during the outpatient clinical encounter that notifies the provider that his or her patient is at risk for stroke due to AF, and that there is no order for anticoagulation. Clinicians who receive the computer alert will have three options: 1) access an order template of United States (US) Food and Drug Administration (FDA)-approved anticoagulation regimens for stroke prevention in AF, 2) follow a link to evidence-based clinical practice guidelines to learn more about stroke prevention in AF, or 3) continue with order entry after providing an explanation for why anticoagulation was not prescribed.
  Interventions: Behavioral: Alert-based computerized decision support
- No Alert (No Intervention): For No Alert cluster sites, no computerized alert notification will be issued to providers.

INTERVENTIONS:
Behavioral: Alert-based computerized decision support — An on-screen electronic alert will be issued during the outpatient clinical encounter that notifies the provider that his or her patient is at risk for stroke due to AF, and that there is no order for anticoagulation. Clinicians who receive the computer alert will have three options: 1) access an order template of FDA-approved anticoagulation regimens for stroke prevention in AF, 2) follow a link to evidence-based clinical practice guidelines to learn more about stroke prevention in AF, or 3) continue with order entry after providing an explanation for why anticoagulation was not prescribed.
  Arms: Alert

SUMMARY:
Atrial fibrillation (AF) is the most preventable cause of stroke. However, despite widely available risk stratification tools, numerous options for oral anticoagulation, and evidence-based practice guidelines, anticoagulation for stroke prevention in AF is consistently under-prescribed. In a pair of observational cohort analyses within the Mass General Brigham (MGB) health system, prescription of anticoagulation for stroke prevention in AF was less frequent in ambulatory clinic patients than in those who were hospitalized at the time of assessment (46.9% vs. 57.2%). Two single academic medical center randomized controlled trials demonstrated success for increasing adherence to guideline recommendations for stroke prevention in AF. To address the feasibility and impact of a computerized decision support (CDS) strategy in the non-tertiary care, community medical center setting, this study will involve a multicenter, cluster-randomized controlled trial of a more sophisticated CDS focused not only on implementation stroke prevention but also on bleeding risk assessment and management.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most preventable cause of stroke. However, despite widely available risk stratification tools, numerous options for oral anticoagulation, and evidence-based practice guidelines, anticoagulation for stroke prevention in AF is consistently under-prescribed. In a pair of observational cohort analyses within the MGB health system, prescription of anticoagulation for stroke prevention in AF was less frequent in ambulatory clinic patients than in those who were hospitalized at the time of assessment (46.9% vs. 57.2%). Implementation science strategies, including computerized decision support (CDS), have been proposed as solutions to improve adherence to guideline recommendations. A previously conducted randomized controlled trial of alert-based CDS in 458 high-risk hospitalized patients with AF who were not being anticoagulated showed that the alert nearly tripled the proportion of hospitalized patients with AF and high-risk of stroke who were prescribed anticoagulation during the hospitalization, at discharge, and at 90 days compared with the control group. CDS in this trial was associated with an 88% reduction in the frequency of stroke or systemic embolic event and 87% reduction in the frequency of myocardial infarction (MI) at 90 days. A subsequent trial demonstrated that clinician-directed, alert-based CDS doubled prescription of antithrombotic therapy in high-risk ambulatory care patients with AF who were not prescribed anticoagulation at the time of randomization. A major lesson from the second trial was the importance that perceived bleeding risk played in the shared decision-making process between clinician and patient. These two trials demonstrated that bleeding risk is the predominant consideration when omitting anticoagulation or choosing to bypass a CDS alert. Clinicians often overestimate bleeding risk compared with objective bleeding risk scores (HAS-BLED).

Both prior trials were executed at a large tertiary-care center in Boston, Massachusetts. The feasibility and impact of an alert-based CDS strategy to improve stroke prevention in AF among ambulatory care patients in the community setting and outside of major tertiary-care centers remains to be determined. To address the feasibility and impact of a CDS strategy in the non-tertiary care, community medical center setting, this study will involve a multicenter, community-based, cluster-randomized controlled trial of a more sophisticated CDS focused not only on implementation stroke prevention but also on bleeding risk assessment and management.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Age ≥ 18 years
* Problem list entry of atrial fibrillation or atrial flutter
* CHA2DS2VASc score ≥ 2 for males
* CHA2DS2VASc score ≥ 3 for females
* No prescription for anticoagulant therapy

Exclusion Criteria:

* Active prescription for anticoagulant therapy
* CHA2DS2VASc score < 2 for males
* CHA2DS2VASc score ≤ 2 for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of prescription of anticoagulation at 90 days in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention at the time of study enrollment | 90 days
  The primary efficacy outcome will be determined by review of the Electronic Health Record (EHR) medication documentation for prescription of anticoagulation by 90 days after enrollment. These data will be collected in the form of a BPA report and then confirmed by independent data abstractors.
Frequency of major bleeding at 6 months from enrollment. | 6 months
  Defined by the ISTH bleeding classification system. These data will be confirmed by independent data abstractors and then independently adjudicated by a blinded 3-physician expert Clinical Events Committee.

SECONDARY OUTCOMES:
Frequency of failure to prescribe anticoagulation because of perceived risk of bleeding in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation at the time of study enrollment and are assigned to the alert group | At 48 hours
  The frequency of this outcome will be compared with that from an earlier study as a historical cohort. This outcome will be determined by review of the EHR.
Frequency of a composite of major adverse cardiovascular events, defined as cerebrovascular accident, systemic embolism, any MI, symptomatic VTE, or all-cause mortality at 6 months from enrollment | 6 months
  The secondary efficacy outcome will be determined by review of the EHR medication documentation. These data will be confirmed by independent data abstractors and then independently adjudicated by a blinded 3-physician expert Clinical Events Committee.

OTHER OUTCOMES:
Frequency of referral for left atrial appendage occlusion among patients with high bleeding risk at 6 months will be reported | 6 months
  Determined by review of the EHR using standardized definition.
Frequency of clinically relevant nonmajor bleeding is defined as overt bleeding not meeting the criteria for major bleeding at 6 months. | 6 months
  Defined by the ISTH bleeding classification system. These data will be confirmed by independent data abstractors and then independently adjudicated by a blinded 3-physician expert Clinical Events Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - St. Elizabeth Health, Edgewood, Kentucky
  - Mass General Brigham, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Piazza G, Hurwitz S, Campia U, Bikdeli B, Lou J, Khairani CD, Bejjani A, Snyder JE, Pfeferman M, Barns B, Rizzo S, Glezer A, Goldhaber SZ. Electronic alerts for ambulatory patients with atrial fibrillation not prescribed anticoagulation: A randomized, controlled trial (AF-ALERT2). Thromb Res. 2023 Jul;227:1-7. doi: 10.1016/j.thromres.2023.05.006. Epub 2023 May 11. PMID 37182298
- [Background] Piazza G, Hurwitz S, Galvin CE, Harrigan L, Baklla S, Hohlfelder B, Carroll B, Landman AB, Emani S, Goldhaber SZ. Alert-based computerized decision support for high-risk hospitalized patients with atrial fibrillation not prescribed anticoagulation: a randomized, controlled trial (AF-ALERT). Eur Heart J. 2020 Mar 7;41(10):1086-1096. doi: 10.1093/eurheartj/ehz385. PMID 31228189